CLINICAL TRIAL: NCT03833479
Title: A Randomized, Open Label, Phase II Trial of Anti-PD1, TSR-042, as Maintenance Therapy for Patients With High-risk Locally Advanced Cervical Cancer After Chemo-radiation
Brief Title: TSR-042 as Maintenance Therapy for Patients With High-risk Locally Advanced Cervical Cancer After Chemo-radiation
Acronym: ATOMICC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: Apices Soluciones S.L. (Industry); GSK/TESARO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICO 78-C (ATOMICC); 2023-510268-11-00 (EU CTIS Number); 2018-002155-15 (EudraCT Number)
Record Dates: First submitted 2019-02-01; First posted 2019-02-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer; Advanced Cancer
Keywords: TSR-042; Anti-PD1; advanced cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No further treatment (Experimental): No further treatment
  Interventions: Other: No Further Treatment
- TSR-042 (Experimental): TSR-042 treatment administered using a 30 -minute IV infusion (with a -5 minute and +15 minute window permitted).
  Interventions: Drug: TSR-042

INTERVENTIONS:
Other: No Further Treatment — No further treatment
  Arms: No further treatment
Drug: TSR-042 — Fixed 500 mg TSR-042 dose Q3W for the first 4 doses followed by a fixed 1000 mg TSR-042 dose Q6W for up to 24 months
  Arms: TSR-042

SUMMARY:
Patients with locally advanced cervical cancer (LACC) despite definitive chemo-radiotherapy, has a poor progression-free survival (PFS) and overall survival (OS). The hypothesis is that the use of TSR-042, checkpoint inhibitor, as consolidation therapy following concurrent chemo-radiation would increase PFS in these patients. The incorporation of immunotherapy after chemo-radiation is one the best scenarios for this approach, since takes advantages of "the ideal microenvironment" created after radiation. In a similar rationale, the phase 3 study that compared the anti-programmed death ligand 1 antibody durvalumab as consolidation therapy with placebo in patients with stage III NSCLC who did not have disease progression after two or more cycles of platinum-based chemoradiotherapy, showed that progression-free survival was significantly longer with durvalumab than with placebo in all sub-groups regardless of response obtained to chemotherapy, namely patients with stable disease (SD) gained the same benefit that patients with partial response (PR). Due to the aforementioned biology of cervical cancer, the proven activity of anti programmed cell death protein 1 (Anti-PD1) agents in metastatic and/or recurrent cervical cancer and the poor PFS and OS in patients with LACC despite definitive chemo-radiotherapy, we consider to analyze the Anti-PD1 agent, TSR-042 as maintenance therapy after concurrent chemo-radiation (CCRT)

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study-specific procedure
2. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
3. Participant must be a female ≥ 18 years of age
4. Life expectancy ≥3 months
5. Participant must have biopsy-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix.
6. Patients must have archival tumor tissue available that is formalin-fixed and paraffin embedded.
7. At diagnosis:

   * Federation of Gynecologists and Obstetricians (FIGO) stages IB2, IIA2, IIB with pelvic lymph node involvement: Biopsy-proven pelvic node involvement, 2 or more positive nodes by magnetic resonance imaging (MRI) or computed tomography (CT) (≥1.5 cm shortest dimension), 2 or more positive nodes by Positron Emission Tomography (PET) (with standardized uptake values (SUV) ≥2.5)
   * FIGO stages IIIA, IIIB, IVA
   * Any FIGO stage with para-aortic lymph node involvement: Biopsy-proven para-aortic node involvement, 1 or more positive nodes by MRI or CT (≥1.5 cm shortest dimension), 1 or more positive pelvic nodes by PET (with SUV ≥ 2.5)
8. Subjects must have received combination chemotherapy and radiotherapy (CCRT) with curative intent. Patients must have received at least 4 doses of weekly cisplatin.
9. Patients must have completed definitive treatment, namely chemo-radiation, up to 12 weeks prior to sign the Informed Consent form.
10. Toxicities resulting from chemo-radiation must resolve to ≤ Grade 1 prior to randomization.
11. Participant must have adequate organ function, defined as follows:

    * Absolute neutrophil count ≥ 1,500/µL
    * Platelets ≥ 100,000/µL
    * Hemoglobin ≥ 9 g/dL
    * Serum creatinine ≤ 1.5× upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using Cockcroft-Gault equation for patients with creatinine levels > 1.5× institutional ULN
    * Total bilirubin ≤ 1.5× ULN OR direct bilirubin ≤ 1× ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN unless liver metastases are present, in which case they must be ≤ 5× ULN
    * International normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
12. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
13. Negative Test Results for Hepatitis
14. Female participant has a negative serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 150 days after the last dose of study treatment, or is of nonchildbearing potential.
15. Participant must agree to not breastfeed during the study or for 150 days after the last dose of study treatment.
16. Male partners must agree to use an adequate method of contraception starting with the first dose of study treatment through 150 days after the last dose of study treatment.
17. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Histological types other than in inclusion criteria, like sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial cancers.
2. FIGO Stage IVB (cancer has spread distantly).
3. Subjects who have undergone a previous hysterectomy defined as removal of the entire uterus or will have a hysterectomy as part of their initial cervical cancer therapy.
4. Has not achieved at least a partial response by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 after completion of CCRT administered with curative intent.
5. Patients previously treated with chemotherapy except when used concurrently with radiation therapy. Patients who have received either concurrent paclitaxel with radiation therapy or carboplatin/paclitaxel as adjuvant therapy are ineligible for the study.
6. Prior treatment with any anti-vascular endothelial growth factor (anti-VEGF) drug, including bevacizumab, CD137 agonists or immune checkpoint blockade therapies, anti-PD1, or anti-PDL1 therapeutic antibodies or anti-CTLA 4.
7. Patients with a concomitant malignancy other than non-melanoma skin cancer.
8. History of autoimmune disease
9. History of idiopathic pulmonary fibrosis, organizing pneumonia , drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
10. History of interstitial lung disease.
11. Active tuberculosis.
12. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
13. Administration of a live, attenuated vaccine within 14 days before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
14. Treatment with systemic immunostimulatory agents within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1.
15. Treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1.
16. Women that are breastfeeding or pregnant.
17. Demonstration of any other disease, neurological or metabolic dysfunction, found upon physical examination or laboratory tests involving a reasonable suspicion of the existence of a disease or condition that contraindicates the use of an experimental drug, or that involves an increased risk to the patient of treatment-related complications.
18. No medical or psychiatric illness that may impede the performance of a systemic or surgical treatment
19. Participant must not be simultaneously enrolled in any interventional clinical trial
20. Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
21. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
22. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
23. Participant must not have a known hypersensitivity to TSR-042 components or excipients.
24. Participant must not have a serious, uncontrolled medical disorder or nonmalignant systemic disease. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
25. Participant must not have known, symptomatic brain or leptomeningeal metastases
26. Patient experienced ≥ Grade 3 immune-related adverse events (AE) with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
27. Participant has a known history of human immunodeficiency virus (type 1 or 2 antibodies).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 134 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 30 months
  Time from the date of randomization to the date of first documentation of disease progression or death due to any cause, whichever occurs first based on investigator assessment using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AEs) | 30 months
  Incidence, nature and severity of adverse events (AEs) assessed by CTCAE version 4.03
Overall survival (OS) | 30 months
  Time from the date of randomization to the date of death due to any cause
Patient reported outcomes (PROs) of health-related quality of life (HRQOL) | 30 months
  Mean changes from baseline score assessed by the Functional Assessment of Cancer Therapy-Cervix (FACT-Cx)
Patient reported outcomes (PROs) of health-related quality of life (HRQOL) | 30 months
  Mean changes from baseline score assessed by EQ -5D-5L.
Patient reported outcomes (PROs) of fatigue | 30 months
  Mean changes from baseline score assessed by the PROMIS-Cancer-Fatigue Short Form 4a.
Patient reported outcomes (PROs) of pain | 30 months
  Mean changes from baseline score assessed by a single item of the Brief Pain Inventory (BPI).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (29):
- Spain (25):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Donostia- Donostia Unibertsitate Ospitalea, Donostia / San Sebastian, Gipuzkoa
  - ICO Girona, Girona, Girona
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - H Vall d'Hebron, Barcelona
  - Hospital Clínic, Barcelona
  - H Reina Sofía Cordoba, Córdoba
  - ICO Hospitalet, Hospitalet Del Llobregat
  - Clinica Universitaria de Navarra, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - H. Parc Taulí, Sabadell
  - Hospital Marqués de Valdecilla, Santander
  - Hospital de Terrassa, Terrassa
- Turkey (Türkiye) (4):
  - Ankara Oncology Training and Research Hospital, Ankara, Anadolu Bölgesi
  - Ankara City Hospital, Ankara, Anadolu Bölgesi
  - Hacettepe University, Ankara, Anadolu Bölgesi
  - Acibadem Maslak Hospital, Istanbul, Sarıyer

REFERENCES:
- [Derived] Garcia-Duran C, Grau F, Villacampa G, Oaknin A. ATOMICC trial: a randomized, open-label, phase II trial of anti-PD1, dostarlimab, as maintenance therapy for patients with high-risk locally advanced cervical cancer after chemoradiation. Int J Gynecol Cancer. 2022 Sep 6;32(9):1196-1200. doi: 10.1136/ijgc-2022-003370. PMID 35444013